CLINICAL TRIAL: NCT02367222
Title: An Observational Retrospective Database Analysis to Estimate the Risk of Multiple Sclerosis Following Vaccination With Arepanrix™ in Manitoba, Canada
Brief Title: A Database Study to Estimate the Risk of Multiple Sclerosis Following Vaccination With Arepanrix™ in Manitoba, Canada
Acronym: H1N1-014VS
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 200405 (H2014:019)
Record Dates: First submitted 2014-12-17; First posted 2015-02-20 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Exposed to Arepanrix™ Cohort: All individuals with Manitoba Immunization Monitoring System (MIMS) record of H1N1 (Arepanrix™) and/or seasonal influenza vaccination during the influenza season 2009/2010 (15 September 2009 to 15 March 2010).
  Interventions: Other: Exposed to Arepanrix™ Cohort
- Unexposed to Arepanrix™ Cohort: All individuals registered with Manitoba Health (MH) during the study period but with no MIMS record for H1N1 (Arepanrix™) and seasonal influenza vaccination during the influenza season 2009/2010 (15 September 2009 to 15 March 2010).
  Interventions: Other: Unexposed to Arepanrix™ Cohort

INTERVENTIONS:
Other: Exposed to Arepanrix™ Cohort — Demographic characteristics such as age, sex, area of residence, socio-economic status; medical history such as comorbidities, immune status, vaccine indication, receipt of other vaccines or medications and frequency of healthcare contacts, as well as information on pregnancy status and pre-existing conditions will be collected..
  Other Names: Database collection and analysis
  Groups: Exposed to Arepanrix™ Cohort
Other: Unexposed to Arepanrix™ Cohort — Demographic characteristics such as age, sex, area of residence, socio-economic status; medical history such as comorbidities, immune status, vaccine indication, receipt of other vaccines or medications and frequency of healthcare contacts, as well as information on pregnancy status and pre-existing conditions will be collected.
  Other Names: Database collection and analysis
  Groups: Unexposed to Arepanrix™ Cohort

SUMMARY:
The purpose of this database study is to assess if Arepanrix™ vaccination during the 2009 pandemic was associated with an increased risk of multiple sclerosis (MS) in Manitoba, Canada.

DETAILED DESCRIPTION:
This observational, retrospective, propensity-score matched cohort study using the Manitoba Immunization Monitoring System (MIMS) and the hospital, physician, and prescription claims databases of the Manitoba Health (MH) Database System will assess if Arepanrix™ vaccination during the 2009 pandemic was associated with an increased risk of multiple sclerosis (MS) and other demyelinating conditions not ultimately leading to a multiple sclerosis diagnosis in Manitoba, Canada.

The data will be collected form the following linked databases:

* Manitoba Health (MH) administrative databases
* Manitoba Immunization Monitoring System (MIMS)
* Manitoba Health Population Registry (MHPR)
* Drug Program Information Network (DPIN)
* Hospital Abstract Database
* The Medical Services database

ELIGIBILITY:
Inclusion Criteria:

* The entire population of Manitoba is considered for inclusion.

Exclusion Criteria:

* Individuals less than or equal to 6 months of age;
* Having less than one year of insurance coverage before the enrolment period;
* Not registered with MH during the enrolment period;
* Physician or hospitalization records indicating a diagnosis of any demyelinating condition between 1971 (earliest year for which information is available) and the index date.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children above 6 months of age (at the time of vaccination) who normally reside in Manitoba, Canada and who had been registered with MH during the study period.
  To ensure sufficient historical data, all participants will be required to have at least one year of insurance coverage before the study period (15 September 2009 to 15 March 2010).
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of MS | 15 September 2009 to 15 March 2010 (up to 6 months)
  During the period of 1 year following administration of Arepanrix™ among an exposed cohort and during an equivalent time period in the unexposed cohort.

SECONDARY OUTCOMES:
Occurrence of MS | 15 September 2009 to 31 December 2012 (up to 39 months)
  From administration of Arepanrix™ until 31 December 2012, among an exposed cohort and during an equivalent time period in the unexposed cohort.
Occurrence of demyelinating events which do not ultimately lead to a diagnosis of MS | 15 September 2009 to 15 March 2010 (up to 3 months)
  During the period of 1 year following administration of Arepanrix™ among an exposed cohort and during an equivalent time period in the unexposed cohort.
Occurrence of demyelinating events which do not ultimately lead to a diagnosis of MS | 15 September 2009 to 31 December 2012 (up to 39 months)
  From administration of Arepanrix™ until 31 December 2012, among an exposed cohort and during an equivalent time period in the unexposed cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Salah Mahmud, MD, PhD, Principal Investigator — Community Health Sciences, University of Manitoba

REFERENCES:
- [Result] Ascherio A, Munger KL, Lunemann JD. The initiation and prevention of multiple sclerosis. Nat Rev Neurol. 2012 Nov 5;8(11):602-12. doi: 10.1038/nrneurol.2012.198. Epub 2012 Oct 9. PMID 23045241
- [Result] Ascherio A, Zhang SM, Hernan MA, Olek MJ, Coplan PM, Brodovicz K, Walker AM. Hepatitis B vaccination and the risk of multiple sclerosis. N Engl J Med. 2001 Feb 1;344(5):327-32. doi: 10.1056/NEJM200102013440502. PMID 11172163
- [Result] Bansil S, Troiano R, Dowling PC, Cook SD. Measles vaccination does not prevent multiple sclerosis. Neuroepidemiology. 1990;9(5):248-54. doi: 10.1159/000110781. PMID 2087249
- [Result] Bardage C, Persson I, Ortqvist A, Bergman U, Ludvigsson JF, Granath F. Neurological and autoimmune disorders after vaccination against pandemic influenza A (H1N1) with a monovalent adjuvanted vaccine: population based cohort study in Stockholm, Sweden. BMJ. 2011 Oct 12;343:d5956. doi: 10.1136/bmj.d5956. PMID 21994316
- [Result] Beck CA, Metz LM, Svenson LW, Patten SB. Regional variation of multiple sclerosis prevalence in Canada. Mult Scler. 2005 Oct;11(5):516-9. doi: 10.1191/1352458505ms1192oa. PMID 16193887
- [Result] Canadian Institute for Health Information (2006). Canadian Classification of Health Interventions (Ottawa, Ontario, Canada).
- [Result] Casetta I, Granieri E, Malagu S, Tola MR, Paolino E, Caniatti LM, Govoni V, Monetti VC, Fainardi E. Environmental risk factors and multiple sclerosis: a community-based, case-control study in the province of Ferrara, Italy. Neuroepidemiology. 1994;13(3):120-8. doi: 10.1159/000110369. PMID 8015665
- [Result] Confavreux C, Suissa S, Saddier P, Bourdes V, Vukusic S; Vaccines in Multiple Sclerosis Study Group. Vaccinations and the risk of relapse in multiple sclerosis. Vaccines in Multiple Sclerosis Study Group. N Engl J Med. 2001 Feb 1;344(5):319-26. doi: 10.1056/NEJM200102013440501. PMID 11172162
- [Result] Cosby SL, McQuaid S, Taylor MJ, Bailey M, Rima BK, Martin SJ, Allen IV. Examination of eight cases of multiple sclerosis and 56 neurological and non-neurological controls for genomic sequences of measles virus, canine distemper virus, simian virus 5 and rubella virus. J Gen Virol. 1989 Aug;70 ( Pt 8):2027-36. doi: 10.1099/0022-1317-70-8-2027. PMID 2769228
- [Result] Cummings P, McKnight B, Greenland S. Matched cohort methods for injury research. Epidemiol Rev. 2003;25:43-50. doi: 10.1093/epirev/mxg002. No abstract available. PMID 12923989
- [Result] Currier RD, Meydrech EF, Currier MM. Measles vaccination has had no effect on the occurrence of multiple sclerosis. Arch Neurol. 1996 Dec;53(12):1216. doi: 10.1001/archneur.1996.00550120018007. No abstract available. PMID 8970447
- [Result] Dean G. How many people in the world have multiple sclerosis? Neuroepidemiology. 1994;13(1-2):1-7. doi: 10.1159/000110351. No abstract available. PMID 8190200
- [Result] DeStefano F, Verstraeten T, Jackson LA, Okoro CA, Benson P, Black SB, Shinefield HR, Mullooly JP, Likosky W, Chen RT; Vaccine Safety Datalink Research Group, National Immunization Program, Centers for Disease Control and Prevention. Vaccinations and risk of central nervous system demyelinating diseases in adults. Arch Neurol. 2003 Apr;60(4):504-9. doi: 10.1001/archneur.60.4.504. PMID 12707063
- [Result] Dublin S, Jackson ML, Nelson JC, Weiss NS, Larson EB, Jackson LA. Statin use and risk of community acquired pneumonia in older people: population based case-control study. BMJ. 2009 Jun 16;338:b2137. doi: 10.1136/bmj.b2137. PMID 19531550
- [Result] Elixhauser A, Steiner C, Harris DR, Coffey RM. Comorbidity measures for use with administrative data. Med Care. 1998 Jan;36(1):8-27. doi: 10.1097/00005650-199801000-00004. PMID 9431328
- [Result] Farez MF, Ysrraelit MC, Fiol M, Correale J. H1N1 vaccination does not increase risk of relapse in multiple sclerosis: a self-controlled case-series study. Mult Scler. 2012 Feb;18(2):254-6. doi: 10.1177/1352458511417253. Epub 2011 Aug 9. No abstract available. PMID 21828198
- [Result] Fedson DS, Wajda A, Nicol JP, Hammond GW, Kaiser DL, Roos LL. Clinical effectiveness of influenza vaccination in Manitoba. JAMA. 1993 Oct 27;270(16):1956-61. PMID 8411553
- [Result] Fleiss J L Levin B, Paik M C. (2003). Statistical Methods for Rates and Proportions (3rd ed.) (Formulas 3.18 &3.19). New York: John Wiley & Sons.
- [Result] Haase AT, Ventura P, Gibbs CJ Jr, Tourtellotte WW. Measles virus nucleotide sequences: detection by hybridization in situ. Science. 1981 May 8;212(4495):672-5. doi: 10.1126/science.7221554.
- [Result] Hammerschlag MR, Ke Z, Lu F, Roblin P, Boman J, Kalman B. Is Chlamydia pneumoniae present in brain lesions of patients with multiple sclerosis? J Clin Microbiol. 2000 Nov;38(11):4274-6. doi: 10.1128/JCM.38.11.4274-4276.2000. PMID 11060110
- [Result] Hardy JR, Holford TR, Hall GC, Bracken MB. Strategies for identifying pregnancies in the automated medical records of the General Practice Research Database. Pharmacoepidemiol Drug Saf. 2004 Nov;13(11):749-59. doi: 10.1002/pds.935. PMID 15386720
- [Result] Humphries KH, Rankin JM, Carere RG, Buller CE, Kiely FM, Spinelli JJ. Co-morbidity data in outcomes research: are clinical data derived from administrative databases a reliable alternative to chart review? J Clin Epidemiol. 2000 Apr;53(4):343-9. doi: 10.1016/s0895-4356(99)00188-2. PMID 10785564
- [Result] Kakalacheva K, Lunemann JD. Environmental triggers of multiple sclerosis. FEBS Lett. 2011 Dec 1;585(23):3724-9. doi: 10.1016/j.febslet.2011.04.006. Epub 2011 Apr 7. PMID 21486562
- [Result] Kelsey JL, Whittemore AS, Evans AS, Thompson WD (1996). Methods in Observational Epidemiology (2nd Edition) (Table 12-15) Oxford University Press.
- [Result] Kozyrskyj AL, Mustard CA. Validation of an electronic, population-based prescription database. Ann Pharmacother. 1998 Nov;32(11):1152-7. doi: 10.1345/aph.18117. PMID 9825079
- [Result] Lix L, Yogendran M, Burchill C, et al., (2006). Defining and Validating Chronic Diseases: An Administrative Data Approach (Winnipeg, Manitoba Centre for Health Policy).
- [Result] Mahmud S, Hammond G, Elliott L, Hilderman T, Kurbis C, Caetano P, Van Caeseele P, Kettner J, Dawood M. Effectiveness of the pandemic H1N1 influenza vaccines against laboratory-confirmed H1N1 infections: population-based case-control study. Vaccine. 2011 Oct 19;29(45):7975-81. doi: 10.1016/j.vaccine.2011.08.068. Epub 2011 Aug 30. PMID 21884747
- [Result] Mahmud SM, Van Caeseele P, Hammond G, Kurbis C, Hilderman T, Elliott L. No association between 2008-09 influenza vaccine and influenza A(H1N1)pdm09 virus infection, Manitoba, Canada, 2009. Emerg Infect Dis. 2012 May;18(5):801-10. doi: 10.3201/eid1805.111596. PMID 22516189
- [Result] Marrie RA, Yu N, Blanchard J, Leung S, Elliott L. The rising prevalence and changing age distribution of multiple sclerosis in Manitoba. Neurology. 2010 Feb 9;74(6):465-71. doi: 10.1212/WNL.0b013e3181cf6ec0. Epub 2010 Jan 13. PMID 20071664
- [Result] Marrie RA. Environmental risk factors in multiple sclerosis aetiology. Lancet Neurol. 2004 Dec;3(12):709-18. doi: 10.1016/S1474-4422(04)00933-0. PMID 15556803
- [Result] MCHP Guidelines for Public and Private Sponsorship of Research Projects Accessing the Population Health Data Repository (2011); http://umanitoba.ca/faculties/medicine/units/community_health_sciences/departmental_units/mchp/protocol/media/Private_Sector_Sponsorship_Guidelines.pdf.
- [Result] McNicholas N, Chataway J. Relapse risk in patients with multiple sclerosis after H1N1 vaccination, with or without seasonal influenza vaccination. J Neurol. 2011 Aug;258(8):1545-7. doi: 10.1007/s00415-011-5944-x. Epub 2011 Feb 19. No abstract available. PMID 21336784
- [Result] Nortvedt MW, Riise T, Myhr KM, Nyland HI. Quality of life in multiple sclerosis: measuring the disease effects more broadly. Neurology. 1999 Sep 22;53(5):1098-103. doi: 10.1212/wnl.53.5.1098. PMID 10496273
- [Result] OpenEpi: Open Source Epidemiologic Statistics for Public Health, Version 3.01, Released April 4 and revised April 6, 2013, http://www.openepi.com/v37/SampleSize/SSPropor.htm.
- [Result] Parsons L S (2001). Reducing bias in a propensity score matched-pair sample using greedy matching techniques. Paper presented at: Proceedings of the Twenty-sixth Annual SAS Users group international conference (SAS Institute, Inc.); pp. 214-26.
- [Result] Persson I, Granath F, Askling J, Ludvigsson JF, Olsson T, Feltelius N. Risks of neurological and immune-related diseases, including narcolepsy, after vaccination with Pandemrix: a population- and registry-based cohort study with over 2 years of follow-up. J Intern Med. 2014 Feb;275(2):172-90. doi: 10.1111/joim.12150. Epub 2013 Nov 10. PMID 24134219
- [Result] Rao SM, Leo GJ, Ellington L, Nauertz T, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. II. Impact on employment and social functioning. Neurology. 1991 May;41(5):692-6. doi: 10.1212/wnl.41.5.692. PMID 1823781
- [Result] Roberts JD, Poffenroth LA, Roos LL, Bebchuk JD, Carter AO. Monitoring childhood immunizations: a Canadian approach. Am J Public Health. 1994 Oct;84(10):1666-8. doi: 10.2105/ajph.84.10.1666. PMID 7943493
- [Result] Roberts JD, Roos LL, Poffenroth LA, Hassard TH, Bebchuk JD, Carter AO, Law B. Surveillance of vaccine-related adverse events in the first year of life: a Manitoba cohort study. J Clin Epidemiol. 1996 Jan;49(1):51-8. doi: 10.1016/0895-4356(95)00522-6. PMID 8598511
- [Result] Roos LL, Mustard CA, Nicol JP, McLerran DF, Malenka DJ, Young TK, Cohen MM. Registries and administrative data: organization and accuracy. Med Care. 1993 Mar;31(3):201-12. doi: 10.1097/00005650-199303000-00002. PMID 8450678
- [Result] Rubin DB. Estimating causal effects from large data sets using propensity scores. Ann Intern Med. 1997 Oct 15;127(8 Pt 2):757-63. doi: 10.7326/0003-4819-127-8_part_2-199710151-00064. PMID 9382394
- [Result] Singh H, Demers AA, Nugent Z, Mahmud SM, Kliewer EV, Bernstein CN. Risk of cervical abnormalities in women with inflammatory bowel disease: a population-based nested case-control study. Gastroenterology. 2009 Feb;136(2):451-8. doi: 10.1053/j.gastro.2008.10.021. Epub 2008 Oct 15. PMID 18996382
- [Result] Singh H, Mahmud SM, Turner D, Xue L, Demers AA, Bernstein CN. Long-term use of statins and risk of colorectal cancer: a population-based study. Am J Gastroenterol. 2009 Dec;104(12):3015-23. doi: 10.1038/ajg.2009.574. Epub 2009 Oct 6. PMID 19809413
- [Result] Skarsgard D, Tonita J. Prostate cancer in Saskatchewan Canada, before and during the PSA era. Cancer Causes Control. 2000 Jan;11(1):79-88. doi: 10.1023/a:1008965617078. PMID 10680732
- [Result] Therneau T M, Grambsch P M (2000). Modeling Survival Data: Extending the Cox Model (New York, Springer).
- [Result] Thompson LH, Mahmud SM, Keynan Y, Blanchard JF, Slater J, Dawood M, Fowke K, Van Caeseele P, Becker M. Serological survey of the novel influenza A H1N1 in inner city Winnipeg, Manitoba, 2009. Can J Infect Dis Med Microbiol. 2012 Summer;23(2):65-70. doi: 10.1155/2012/484693. PMID 23730311
- [Result] Vrethem M, Malmgren K, Lindh J. A patient with both narcolepsy and multiple sclerosis in association with Pandemrix vaccination. J Neurol Sci. 2012 Oct 15;321(1-2):89-91. doi: 10.1016/j.jns.2012.07.025. Epub 2012 Jul 28. PMID 22841884
- [Result] WHO Collaborating Centre for Drug Statistics Methodology (2002). ATC Index With DDDs (WHO, Oslo, Norway,).
- [Result] Bramer GR. International statistical classification of diseases and related health problems. Tenth revision. World Health Stat Q. 1988;41(1):32-6. PMID 3376487
- [Result] Robinson JR, Young TK, Roos LL, Gelskey DE. Estimating the burden of disease. Comparing administrative data and self-reports. Med Care. 1997 Sep;35(9):932-47. doi: 10.1097/00005650-199709000-00006. PMID 9298082
- [Result] Zarychanski R, Stuart TL, Kumar A, Doucette S, Elliott L, Kettner J, Plummer F. Correlates of severe disease in patients with 2009 pandemic influenza (H1N1) virus infection. CMAJ. 2010 Feb 23;182(3):257-64. doi: 10.1503/cmaj.091884. Epub 2010 Jan 21. PMID 20093297
- [Result] Zorzon M, Zivadinov R, Nasuelli D, Dolfini P, Bosco A, Bratina A, Tommasi MA, Locatelli L, Cazzato G. Risk factors of multiple sclerosis: a case-control study. Neurol Sci. 2003 Nov;24(4):242-7. doi: 10.1007/s10072-003-0147-6. PMID 14658040